CLINICAL TRIAL: NCT06875336
Title: A Multicentric Cohort and Biomarker Study for Improved Care of Patients with Extrapulmonary Tuberculosis
Acronym: mEX-TB
Status: Recruiting | Type: Observational
Sponsor: University of Cologne (Other)
Collaborators: University Hospital, Bonn (Other); Research Center Borstel (Other); Johann Wolfgang Goethe University Hospital (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University Hospital Heidelberg (Other); Helmholtz Zentrum München (Industry); University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Isabelle Suarez, Attending Physician, University of Cologne
Other Study IDs: TTU 02.913_00
Record Dates: First submitted 2023-05-12; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Extrapulmonary Tuberculosis
Keywords: extrapulmonary tuberculosis; biomarker; cohort study
MeSH Terms: conditions — Tuberculosis, Extrapulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum urine heparin blood PAXgene blood sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with extrapulmonary tuberculosis: During the visits routine clinical and laboratory parameters (assessment of symptoms e.g. pain, weight gain, blood count, liver enzymes, renal parameters, vitamin D levels, CRP etc.), radiographic imaging (ultrasound, CT scan or MRI) and drug specific parameters (dose, interval, adverse events) are documented. Moreover, 3 sputum specimens (on 3 different days) and 1 urine specimen are collected initially for microscopy, PCR and culture through in-house microbiology departments.
  A paper case record form (CRF) will be used to collect patient data, which will be then transferred to an electronic database by local study personnel.
  At each time-point a series of additional specimens, consisting of serum, urine, heparin blood, and PAXgene blood for RNA will be collected and stored. If M. tuberculosis can be cultivated, strains will be stored for genotyping and whole genome sequencing. Serum biomarkers will be tested using commercially available kits.
  Interventions: Diagnostic Test: biomarker analysis

INTERVENTIONS:
Diagnostic Test: biomarker analysis — PAXgene blood for RNA will be collected and stored. Results from these additional examinations are not included in the treatment monitoring of the patient concerned. If M. tuberculosis can be cultivated, strains will be stored for genotyping and whole genome sequencing. Serum biomarkers will be tested using commercially available kits.
  In addition, TAM-TB assays will be performed from samples stored at each time-point. For this purpose, PBMCs will be collected and frozen using well-established protocols.

SUMMARY:
This is a prospective, multicenter, observational study (mEX-TB study) of patients with extrapulmonary tuberculosis (EPTB). Adult patients newly diagnosed with EPTB will prospectively be enrolled into the study. Clinical data will be collected using standardized questionnaires over the whole treatment period for each individual. Additionally, body fluids (blood, urine) will be collected and stored in a central biobank. Biomarkers in EPTB patients will be analyzed during the course of therapy and correlated with clinical data. In addition, a healthy control group will be added, to be used primarily as technical controls for complex laboratory procedures such as RNA-seq and T-cell based assays.

DETAILED DESCRIPTION:
Background: According to the World Health Organization (WHO), 10 million people fell ill with tuberculosis (TB) in 2019, and 1.4 million people died from this disease. Among infectious agents, Mycobacterium tuberculosis (Mtb) remains the major cause of mortality and morbidity worldwide. Control of the disease is increasingly complicated due to growing numbers of infections with multi-drug resistant strains. In Germany, we witnessed a sharp increase of new cases (7.3 cases per 100,000) in 2015. From 2016 to 2017 the incidence decreased, while the numbers in 2018 (5,429 reported TB cases; 6.5 cases per 100,000) kept almost unchanged. Migrants from high incidence areas account for the majority of all TB patients (67,1% in 2019). While pulmonary TB (PTB) is the most common manifestation, any other organ can be involved. Extrapulmonary TB (EPTB) constitutes for 27,8% (1,321) of all cases in Germany. While the overall incidence of TB is decreasing in industrialized countries, the proportion of EPTB has been constantly increasing in Germany and other European countries. The reasons for this are not fully understood. An extensive retrospective study performed in China showed a significantly higher proportion of multi-drug resistant TB among patients with EPTB than among patients with PTB. This clearly highlights the need for improved EPTB control measures in order to avoid the development of drug resistance and to achieve the goal of TB eradication on a national and international level (e.g. WHO End-TB-strategy) which is further challenged by the SARS-CoV-2 pandemic. The mEX-TB project focuses on EPTB with the main goal of optimizing clinical management of EPTB patients. A prospective clinical cohort of EPTB will be established, involving multiple researchers and clinical sites (Frankfurt, Heidelberg, Borstel, Hamburg, Bonn, Cologne), which will enable us to conduct detailed clinical and translational studies addressing this disease entity.

Description:

Study population, research design and research methods Adult patients newly diagnosed with EPTB (N=150) will prospectively be enrolled into the study. PTB patients (N=30) will also be included and serve as a control group to test the technical feasibility. In addition, a healthy control group (N=30) will be added, mainly to address aim 1. Clinical data will be collected using standardized questionnaires over the whole treatment period for each individual.

Additionally, body fluids (blood, urine) will be collected and stored in a central biobank (Cologne). However, not all contributing centers will be able to provide high quality peripheral blood mononuclear cells (PBMCs) for storage. In order not to lose patients with incomplete sample collections, the cohort study will have several strata:

1. EPTB patients (N=100) with clinical data (e.g. weight gain, imaging results etc.) and a full collection of bio samples (routine laboratory parameters, peripheral blood mononuclear cells (PBMCs), PAXgene RNA/DNA tubes for gene signatures, absolute and relative CD4/CD8 cell count, Vitamin D (25(OH)D), urine, plasma)
2. EPTB patients (N=50) with clinical data (e.g. weight gain, imaging results, microbiology results etc.) plus/minus a partial collection of bio samples (e.g. routine laboratory results, Vitamin D (25(OH)D), PAXgene, plasma)
3. Healthy controls (N=30) and a full collection of bio samples as described for stratum 1 at one timepoint.

Data collection Pseudonymized clinical and laboratory data will be recorded at the following time points: diagnosis/ treatment initiation (day 0 / +/- 7 days); 4 weeks post treatment initiation (+/- 7 days); 3 months post treatment initiation (+/- 7 days); 6 months post treatment initiation (+/- 7 days); 3 months post end of treatment (+/- 7 days). In patients requiring treatment of more than 6 months (i.e. multi-drug resistant TB, disseminated TB etc.) data will be collected regularly until end of treatment. Pseudonymization of patient data and acquisition of biomaterial is performed through a patient ID-generator. A paper case report form (CRF) will be used to collect patient data. The CRF data will be then transferred to an electronic database.

Outcome:

Laboratory based biomarkers for assessing treatment responses similar to sputum conversion used for PTB are not available in most cases of EPTB. Unspecific inflammation markers such as C-reactive protein (CRP) can be utilized to assess early treatment response. We will systematically and longitudinally assess radiologic parameters (lesion size in CT, ultrasonography or MRI), laboratory findings and clinical signs (e.g. weight gain, less pain, absence of fever etc.). We will then exploit response algorithms specifically evaluated for EPTB patients initiating anti-TB treatment. A combination of three clinical parameters will be used 1) improvement in reported symptoms 2) weight gain (any weight gain or ≥ 5% weight gain) 3) regression of lymph node swelling, pleural or peritoneal effusion or other local findings, during and after treatment. A combination of these parameters predicts favorable or unfavorable outcome early during the treatment process.

Aims:

Our aim is to assess the treatment response using these parameters, supported by two independent clinicians and experts in the field (blind review). Data will be correlated with blood based biomarker findings described below. The main objectives of this study are the development of EPTB specific biomarkers for improved EPTB diagnostics and assessment of treatment responses by correlating immunological and blood based parameters and signatures with clinical features at baseline and longitudinally. For this purpose, our biomarker study will focus on two major aims:

Study aim I: Evaluation of blood biomarkers as diagnostic tools for EPTB Sputum or lung fluid based laboratory diagnostics as performed with PTB is not possible in most cases of EPTB. Blood based biomarkers are required.

* We will focus on two approaches: 1) blood derived gene expression signatures associated with tuberculosis; 2) T-cell based assays (e.g. TAM-TB assay).
* For this aim, we will first investigate markers that have already been analyzed in PTB patients. We will also be able to investigate EPTB specific markers in an unbiased fashion if necessary.

Study aim II: Evaluation of blood biomarkers predicting treatment response or failure and cure in EPTB

* Predicting cure or the risk of treatment failure is crucial for the management of EPTB. Various outcome definitions for PTB are based on culture and smear results which is not applicable in EPTB. Our aim is to correlate blood based biomarkers with the treatment response which we will assess with well-defined clinical parameters.
* For this aim we will continue with our evaluation of plasma IP-10 as a simple and cost-effective treatment response marker. Additional plasma-based markers have been described in our proposal. More complex markers/signatures (gene expression via RNA-seq and T-cell response based) will be applied using technical approaches similar to the ones exploited in Aim 1. We will primarily focus on signatures that have already been evaluated for PTB. The overarching goal of this unique multicenter cohort of patients with EPTB is the development.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Isolation of Mycobacterium tuberculosis complex from a bodily secretion or tissue by

   1. PCR
   2. culture or a presumptive clinical diagnosis based on epidemiologic exposure in combination with physical findings, radiographic findings and/or histopathology
3. Patients with extrapulmonary TB

   * pleura
   * lymph nodes
   * bones and joints
   * larynx
   * pericardial
   * parotid gland
   * abdominal sites
   * kidneys
   * genitourinary tract
   * disseminated (miliary) TB
   * other than pulmonary TB
4. In the case of pulmonary and extrapulmonary involvement, the leading manifestation, clinically and radiographically, must be extrapulmonary.
5. Written informed consent provided prior to inclusion

Exclusion Criteria:

* 1. Age <18 years 2. Patient with any social or logistical condition which, as anticipated by the investigator, may interfere with the conduct of the study, such as incapacity to well understand the study content and procedure (in case of any language barriers, a translator may be involved), not willing to collaborate, or anticipated inability to finish study due to physical weakness 3. Dependencies towards the study team (e.g. family members, employees of the same department) 4. Pregnant women 5. Patient in custodianship or guardianship 6. Leading pulmonary manifestation 7. Solitary CNS tuberculosis Patients may take part in other clinical studies and trials, as long as there is no conflict with the inclusion or exclusion criteria of the mEX-TB study and the protocol of the other study or trial does not conflict with the means of data and sample collection and publication of this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are regular patients at the University Hospital of Cologne
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of blood biomarkers as diagnostic tools for EPTB (gene expression via RNA-seq and T-cell response based) | two years
  There is limited research on extrapumonary tuberculosis. In particular, it is difficult to establish the diagnosis. Therefore, one aim of this study is to investigate biomarkers (gene expression via RNA-seq and T-cell response based) that have been shown to be effective for pumonal tuberculosis also for extrapulmonary tuberculosis.
Evaluation of blood biomarkers to predict treatment response or failure, and cure in EPTB | two years
  There is limited research on extrapumonary tuberculosis. In particular, treatment duration is difficult to estimate. Therefore, one aim of this study is to investigate biomarkers (gene expression via RNA-seq and T-cell response based) that have been shown to be useful for pulmonary tuberculosis also for extrapulmonary tuberculosis.

SECONDARY OUTCOMES:
Evaluation of clinical data to identify risk factors for dissemination of the disease (limited vs severe disease) | two years
  The clinical picture of extrapulmonary tuberculosis is very heterogeneous and it is still not clear which factors lead to the development of lymph node tuberculosis in some patients and disseminated disease in others. Using the clinical cohort, the disease pattern will be described more precisely.
Influence of former refugee experience on the spread of the disease | two years
  The clinical picture of extrapulmonary tuberculosis is very heterogeneous and it is still not clear which factors lead to the development of lymph node tuberculosis in some patients and disseminated disease in others. Using the clinical cohort, the disease pattern will be described more precisely.
Proportion and description of paradoxical reaction and identifying biomarkers predicting occurrence of paradoxical reactions (e.g. IP-10) | two years
  Risk factors for the occurrence of paradoxical reactions will be identified by analyzing clinical data.

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - University Hospital Bonn, Bonn
  - Research Center Borstel, Borstel
  - University Hospital of Cologne, Cologne
  - University Hospital Frankfurt, Frankfurt
  - University Hospital Hamburg, Hamburg
  - University Hospital Heidelberg, Heidelberg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fortun J, Martin-Davila P, Gomez-Mampaso E, Gonzalez-Garcia A, Barbolla I, Gomez-Garcia I, Wikman P, Ortiz J, Navas E, Cuartero C, Gijon D, Moreno S. Extra-pulmonary tuberculosis: differential aspects and role of 16S-rRNA in urine. Int J Tuberc Lung Dis. 2014 Apr;18(4):478-85. doi: 10.5588/ijtld.13.0555. PMID 24670706
- [Background] Gonzalez-Garcia A, Fortun J, Elorza Navas E, Martin-Davila P, Tato M, Gomez-Mampaso E, Moreno S. The changing epidemiology of tuberculosis in a Spanish tertiary hospital (1995-2013). Medicine (Baltimore). 2017 Jun;96(26):e7219. doi: 10.1097/MD.0000000000007219. PMID 28658113
- [Background] Grab J, Suarez I, van Gumpel E, Winter S, Schreiber F, Esser A, Holscher C, Fritsch M, Herb M, Schramm M, Wachsmuth L, Pallasch C, Pasparakis M, Kashkar H, Rybniker J. Corticosteroids inhibit Mycobacterium tuberculosis-induced necrotic host cell death by abrogating mitochondrial membrane permeability transition. Nat Commun. 2019 Feb 8;10(1):688. doi: 10.1038/s41467-019-08405-9. PMID 30737374
- [Background] Graham SM, Cuevas LE, Jean-Philippe P, Browning R, Casenghi M, Detjen AK, Gnanashanmugam D, Hesseling AC, Kampmann B, Mandalakas A, Marais BJ, Schito M, Spiegel HM, Starke JR, Worrell C, Zar HJ. Clinical Case Definitions for Classification of Intrathoracic Tuberculosis in Children: An Update. Clin Infect Dis. 2015 Oct 15;61Suppl 3(Suppl 3):S179-87. doi: 10.1093/cid/civ581. PMID 26409281
- [Background] Mihret A, Bekele Y, Bobosha K, Kidd M, Aseffa A, Howe R, Walzl G. Plasma cytokines and chemokines differentiate between active disease and non-active tuberculosis infection. J Infect. 2013 Apr;66(4):357-65. doi: 10.1016/j.jinf.2012.11.005. Epub 2012 Nov 20. PMID 23178506
- [Background] Mulenga H, Zauchenberger CZ, Bunyasi EW, Mbandi SK, Mendelsohn SC, Kagina B, Penn-Nicholson A, Scriba TJ, Hatherill M. Performance of diagnostic and predictive host blood transcriptomic signatures for Tuberculosis disease: A systematic review and meta-analysis. PLoS One. 2020 Aug 21;15(8):e0237574. doi: 10.1371/journal.pone.0237574. eCollection 2020. PMID 32822359
- [Background] Odone A, Tillmann T, Sandgren A, Williams G, Rechel B, Ingleby D, Noori T, Mladovsky P, McKee M. Tuberculosis among migrant populations in the European Union and the European Economic Area. Eur J Public Health. 2015 Jun;25(3):506-12. doi: 10.1093/eurpub/cku208. Epub 2014 Dec 13. PMID 25500265
- [Background] Pai M, Nicol MP, Boehme CC. Tuberculosis Diagnostics: State of the Art and Future Directions. Microbiol Spectr. 2016 Oct;4(5). doi: 10.1128/microbiolspec.TBTB2-0019-2016. PMID 27763258
- [Background] Pang Y, An J, Shu W, Huo F, Chu N, Gao M, Qin S, Huang H, Chen X, Xu S. Epidemiology of Extrapulmonary Tuberculosis among Inpatients, China, 2008-2017. Emerg Infect Dis. 2019 Mar;25(3):457-464. doi: 10.3201/eid2503.180572. PMID 30789144
- [Background] Schaberg T, Bauer T, Brinkmann F, Diel R, Feiterna-Sperling C, Haas W, Hartmann P, Hauer B, Heyckendorf J, Lange C, Nienhaus A, Otto-Knapp R, Priwitzer M, Richter E, Rumetshofer R, Schenkel K, Schoch OD, Schonfeld N, Stahlmann R. [Tuberculosis Guideline for Adults - Guideline for Diagnosis and Treatment of Tuberculosis including LTBI Testing and Treatment of the German Central Committee (DZK) and the German Respiratory Society (DGP)]. Pneumologie. 2017 Jun;71(6):325-397. doi: 10.1055/s-0043-105954. Epub 2017 Jun 26. German. PMID 28651293
- [Background] Suarez I, Maria Funger S, Jung N, Lehmann C, Reimer RP, Mehrkens D, Bunte A, Plum G, Jaspers N, Schmidt M, Fatkenheuer G, Rybniker J. Severe disseminated tuberculosis in HIV-negative refugees. Lancet Infect Dis. 2019 Oct;19(10):e352-e359. doi: 10.1016/S1473-3099(19)30162-8. Epub 2019 Jun 7. PMID 31182290
- [Background] Paul G, Wesselmann J, Adzic D, Malin JJ, Suarez I, Priesner V, Kummerle T, Wyen C, Jung N, van Bremen K, Schlabe S, Wasmuth JC, Boesecke C, Fatkenheuer G, Rockstroh J, Schwarze-Zander C, Lehmann C. Predictors of serofast state after treatment for early syphilis in HIV-infected patients. HIV Med. 2021 Mar;22(3):165-171. doi: 10.1111/hiv.12985. Epub 2020 Oct 30. PMID 33128333
- [Background] Warnat-Herresthal S, Schultze H, Shastry KL, Manamohan S, Mukherjee S, Garg V, Sarveswara R, Handler K, Pickkers P, Aziz NA, Ktena S, Tran F, Bitzer M, Ossowski S, Casadei N, Herr C, Petersheim D, Behrends U, Kern F, Fehlmann T, Schommers P, Lehmann C, Augustin M, Rybniker J, Altmuller J, Mishra N, Bernardes JP, Kramer B, Bonaguro L, Schulte-Schrepping J, De Domenico E, Siever C, Kraut M, Desai M, Monnet B, Saridaki M, Siegel CM, Drews A, Nuesch-Germano M, Theis H, Heyckendorf J, Schreiber S, Kim-Hellmuth S; COVID-19 Aachen Study (COVAS); Nattermann J, Skowasch D, Kurth I, Keller A, Bals R, Nurnberg P, Riess O, Rosenstiel P, Netea MG, Theis F, Mukherjee S, Backes M, Aschenbrenner AC, Ulas T; Deutsche COVID-19 Omics Initiative (DeCOI); Breteler MMB, Giamarellos-Bourboulis EJ, Kox M, Becker M, Cheran S, Woodacre MS, Goh EL, Schultze JL. Swarm Learning for decentralized and confidential clinical machine learning. Nature. 2021 Jun;594(7862):265-270. doi: 10.1038/s41586-021-03583-3. Epub 2021 May 26. PMID 34040261
- [Background] Treatment of Tuberculosis: Guidelines. 4th edition. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK138748/ PMID 23741786
- [Background] WHO consolidated guidelines on tuberculosis: Module 4: Treatment - Drug-resistant tuberculosis treatment [Internet]. Geneva: World Health Organization; 2020. Available from http://www.ncbi.nlm.nih.gov/books/NBK558570/ PMID 32603040
- [Background] Chakaya J, Petersen E, Nantanda R, Mungai BN, Migliori GB, Amanullah F, Lungu P, Ntoumi F, Kumarasamy N, Maeurer M, Zumla A. The WHO Global Tuberculosis 2021 Report - not so good news and turning the tide back to End TB. Int J Infect Dis. 2022 Nov;124 Suppl 1:S26-S29. doi: 10.1016/j.ijid.2022.03.011. Epub 2022 Mar 20. PMID 35321845
- [Background] Chakaya J, Khan M, Ntoumi F, Aklillu E, Fatima R, Mwaba P, Kapata N, Mfinanga S, Hasnain SE, Katoto PDMC, Bulabula ANH, Sam-Agudu NA, Nachega JB, Tiberi S, McHugh TD, Abubakar I, Zumla A. Global Tuberculosis Report 2020 - Reflections on the Global TB burden, treatment and prevention efforts. Int J Infect Dis. 2021 Dec;113 Suppl 1(Suppl 1):S7-S12. doi: 10.1016/j.ijid.2021.02.107. Epub 2021 Mar 11. PMID 33716195